CLINICAL TRIAL: NCT07042958
Title: Evaluation of Customized Zirconia Membrane in Direct Sinus Lifting With Simultaneous Implant Placement: (Randomized Control Trial)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Aliaa Shaban Mohamed, Aliaa Shaban Mohamed, Fayoum University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: the number obtain at end study
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Sinus Lifting
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental)
  Interventions: Procedure: zirconia membrane
- control group): (Experimental)
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: zirconia membrane — Patients with atrophic maxilla will undergo a direct sinus lift procedure, utilizing a customized zirconia membrane for tenting, along with simultaneous implant placement.
  Arms: Study group
Procedure: control group — Patients with atrophic maxilla will undergo a direct sinus lift procedure, using tenting with simultaneous implant placement.
  Arms: control group):

SUMMARY:
Modern dental implantology offers solutions for patients with edentulism in the maxillary arch, where sinus pneumatization and alveolar ridge atrophy are common. This requires sinus floor elevation and bone grafting for implant placement. Techniques like the lateral window approach and osteotome-mediated sinus floor elevation aim to achieve the necessary vertical bone height for implants. Autogenous bone grafts have been the gold standard but have limitations like donor site morbidity and graft volume loss, leading to the exploration of alternatives. Membranes, such as resorbable collagen or titanium-reinforced materials, are commonly used in these procedures but have limitations related to customization, cost, and failure rates.Recent studies have suggested that placing implants directly into the sinus without grafting material can stimulate bone formation, leveraging blood clots to activate bone-forming cells. Zirconia, a ceramic material known for its bioinertness and mechanical strength, is being explored for its potential in sinus lift procedures. Customized 3D zirconia membranes may offer a solution to enhance bone formation and soft tissue integration during sinus lifts.This study aims to evaluate the effect of using customized zirconia membranes in sinus lift procedures with simultaneous implant placement, comparing bone height outcomes with conventional sinus lifts without membranes

DETAILED DESCRIPTION:
Modern dental implantology offers solutions for patients with edentulism in the maxillary arch, where sinus pneumatization and alveolar ridge atrophy are common. This requires sinus floor elevation and bone grafting for implant placement. Techniques like the lateral window approach and osteotome-mediated sinus floor elevation aim to achieve the necessary vertical bone height for implants. Autogenous bone grafts have been the gold standard but have limitations like donor site morbidity and graft volume loss, leading to the exploration of alternatives. Membranes, such as resorbable collagen or titanium-reinforced materials, are commonly used in these procedures but have limitations related to customization, cost, and failure rates.Recent studies have suggested that placing implants directly into the sinus without grafting material can stimulate bone formation, leveraging blood clots to activate bone-forming cells. Zirconia, a ceramic material known for its bioinertness and mechanical strength, is being explored for its potential in sinus lift procedures. Customized 3D zirconia membranes may offer a solution to enhance bone formation and soft tissue integration during sinus lifts.This study aims to evaluate the effect of using customized zirconia membranes in sinus lift procedures with simultaneous implant placement, comparing bone height outcomes with conventional sinus lifts without membranes Objectives: The study will assess bone height after sinus lift with customized zirconia membranes versus conventional sinus lift without membranes.

Methods: A randomized clinical trial will compare two groups: one using a customized zirconia membrane and implant placement, and the other receiving the procedure without the membrane. Preoperative assessments will include CBCT and CAD-guided planning, followed by implantation and postoperative monitoring to assess bone height, density, and implant stability.

ELIGIBILITY:
Patient will be selected according to certain inclusion and exclusion criteria:

1. Inclusion criteria Patient with Atrophic posterior maxilla and remaining bone height less than 6 mm.

I. ASA physical status I and II. II. Patient with healthy maxillary sinus free from any pathology. III. The edentulous ridges are covered with optimal thickness of Mucoperiosteum with no signs of inflammation, ulceration or scar tissue.

IV. Occlusion showed sufficient inter arch space for future prosthesis.

Exclusion Criteria:

General contraindications to implant surgery. I. Untreated gingivitis, periodontitis. II. Patient with maxillary sinusitis. III. Smoker patient. IV. Patient with parafunctional habits. V. Subjected to irradiation in the head and neck area less than 1 year before implantation.

VI. Pregnant or nursing.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Gained bone height | 6month